CLINICAL TRIAL: NCT04772768
Title: Patients With Prior Coronary Artery Bypass Graft Surgery Evaluated for Saphenous VeIn grAft DysfUnction and Progression of Coronary arTery Disease
Brief Title: Prior CABG Patients Evaluated for Saphenous VeIn grAft DysfUnction and Progression of Coronary arTery Disease
Acronym: VIADUCT
Status: Recruiting | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Paul Knaapen, Principle investigator, MD, PhD, Professor of Cardiac Intervention and Imaging, Amsterdam UMC, location VUmc
Other Study IDs: Amsterdam UMC 2019.457
Record Dates: First submitted 2021-02-22; First posted 2021-02-26 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Recurrent Angina After Coronary Artery Bypass Graft; Graft Failure; Coronary Artery Disease Progression
Keywords: Coronary Artery Bypass Grafting; Recurrent angina; Saphenous vein graft dysfunction; Advanced coronary artery disease
MeSH Terms: conditions — Angina Pectoris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multi-center, observational cohort study including patients with prior coronary artery bypass grafting (CABG) and ≥1 saphenous vein grafts (SVG) presenting with recurrent ischemic symptoms. Objective: to investigate the clinical outcomes in patients with prior CABG evaluated for bypass graft failure and progression of native coronary artery disease (CAD). Follow-up will be collected through national registry databases, electronic medical patient records and standardized telephonic assessment at 3 and 5 years follow-up.

DETAILED DESCRIPTION:
Despite advances in secondary prevention, a wide variety of vascular grafts available, and evolving surgical techniques, long-term efficacy of CABG is hampered by bypass graft failure and native CAD progression. Therefore, patients with prior CABG often present with recurrent ischemic symptoms. Indeed, many prior CABG patients undergo repeat cardiac catheterization and require subsequent revascularization therapy. The clinical evaluation and diagnostic work-up of patients with recurrent angina after CABG is challenging. Patients with previous CABG are generally older, have a higher prevalence of cardiac risk factors and comorbidities, more extensive CAD, and complex atherosclerotic lesion morphology. Furthermore, current guideline recommendations on patient management are limited since post-CABG patients have often been underrepresented or excluded in large diagnostic and revascularization trials. This registry will include patients presenting with recurrent ischemic symptoms with a history of CABG and ≥1 SVGs that are referred to the Amsterdam University Medical Centers. Patients will be eligible for inclusion in the VIADUCT registry after consideration of in- and exclusion criteria. Subsequently, patients will be approached for study participation. Patients are free to refuse or to withdraw from participation in the registry at any moment. The primary objective is to investigate clinical outcomes in patients with recurrent symptoms who are evaluated for bypass graft failure and native CAD progression. In addition, results from non-invasive and invasive diagnostic tools that are used during clinical work-up to assess graft patency, the hemodynamic significance of native CAD progression, left ventricular function, and myocardial viability will be collected. We aim to evaluate the value of such tools to guide optimal repeat revascularization strategy.

ELIGIBILITY:
Inclusion Criteria:

* Prior coronary artery bypass grafting
* One or more saphenous vein grafts
* Recurrent angina symptoms

Exclusion Criteria:

* <18 years of age
* ≥ 90 years of age
* Cardiogenic shock
* Pregnancy
* Failure to provide informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with recurrent angina symptoms and a cardiac history of CABG with one or more saphenous vein grafts evaluated for saphenous vein graft dysfunction and progression of coronary artery disease in the Amsterdam University Medical Centers, Department of Cardiology
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-08-23 (Actual); Primary Completion 2024-07-23 (Estimated); Study Completion 2029-07-23 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events (MACE) | 3 year follow-up
  The total number and specification of major adverse cardiac events (all-cause mortality, non-fatal myocardial infarction, or clinically driven repeat revascularization)
Saphenous vein graft failure | At the time of referral and during subsequent 3 and 5 years follow-up
  Failure rate and duration of graft patency following prior CABG procedure

SECONDARY OUTCOMES:
Major Adverse Cardiac Events | 3 and 5 years follow-up
  Components of MACE (all-cause mortality, non-fatal myocardial infarction, or clinically driven repeat revascularization)
Procedural success and mortality in patients who underwent percutaneous coronary intervention of a saphenous vein graft | In hospital and during subsequent 3 and 5 years follow-up
  Procedural success defined by technical success and no major in-hospital complications (mortality, stroke, myocardial infarction, tamponade requiring centesis, emergency CABG/PCI, acute kidney failure requiring dialysis, vascular access site complication or major bleeding requiring transfusion or surgery)
Procedural success and mortality in patients who underwent percutaneous coronary intervention of a (bypassed) native coronary artery | In hospital and during subsequent 3 and 5 years follow-up
  Procedural success defined by technical success and no major in-hospital complications (mortality, stroke, myocardial infarction, tamponade requiring centesis, emergency CABG/PCI, acute kidney failure requiring dialysis, vascular access site complication or major bleeding requiring transfusion or surgery)
Quality of life assessed by the Canadian Cardiovascular Society (CCS) Grading Scale | At baseline and during subsequent 3 and 5 years follow-up
  Canadian Cardiovascular Society (CCS) Grading Scale measures whether patient have angina pectoris complaints, and to what extent patients experienced this. It uses a scale of 1-4 where 1 means angina pectoris (chest pain) only occurs with strenuous, rapid or prolonged exertion, and 4 means angina is present during little physical effort or even during rest.
Quality of life assessed by Rose dyspnea scale questionnaire (RDS) | At baseline and during subsequent 3 and 5 years follow-up
  Rose dyspnea scale questionnaire (RDS) measures dyspnea complaints, or shortness of breath. It consists of 4 questions about dyspnea complaints in the everyday life of patients. For every patient, a score is compiled of the highest limitation in daily life, resulting in a score of 0-4, where 0 means no dyspnea complaints and 4 means the patient has complaints during no or minimal physical effort.
Composite score of quality of life | At baseline and during subsequent 3 and 5 years follow-up
  Composite of all quality of life questionnaires, where all outcomes are summed to provide a total score

CONTACTS AND LOCATIONS:
Overall Officials: Paul Knaapen, Professor, Principal Investigator — Amsterdam University Medical Centers, Department of Cardiology
Locations (1):
- Amsterdam University Medical Centers, Department of Cardiology, Amsterdam, Netherlands

REFERENCES:
- [Derived] Hoek R, de Winter RW, Peters RT, Somsen YBO, van Diemen PA, Jukema RA, Twisk JW, Verouden NJ, den Hartog AW, Raijmakers PG, Nap A, Danad I, Knaapen P. Comparison of Fractional Flow Reserve and Myocardial Perfusion Imaging in Saphenous Vein Grafts. Catheter Cardiovasc Interv. 2025 May;105(6):1365-1374. doi: 10.1002/ccd.31467. Epub 2025 Feb 24. PMID 39991799